CLINICAL TRIAL: NCT04591912
Title: Randomized Controlled Trial of the Peer-Delivered "Mind. Body. Voice." Eating Disorder Prevention Program Among High School Women - Remote
Brief Title: The Peer-Delivered "Mind. Body. Voice." Program for High School Women (Mbv) - Remote
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Sona Dimidjian, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0007-03
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Eating Disorders in Adolescence
Keywords: Eating disorder prevention; Peer delivery; Female; Adolescence
MeSH Terms: interventions — Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mind. body. voice. (Experimental): The 10-week mind. body. voice. program.
  Interventions: Behavioral: mind. body. voice
- Control (No Intervention): Assessment-only control

INTERVENTIONS:
Behavioral: mind. body. voice — The mbv program consists of 10 weekly sessions that include a variety of practices, including: cognitive dissonance exercises, contemplative practices, guided discussion and community building.
  Other Names: Healthy Body, Mind, and Voice
  Arms: mind. body. voice.

SUMMARY:
This study will evaluate the impact of a program (called mind. body. voice. or "mbv") that was collaboratively designed by youth, educators, and researchers, informed by the Body Project (Becker et al., 2013; Stice et al., 2019), Youth Participatory Action Research, an extended co-design process, and previous iterations of the mbv program. The study evaluates the impact of the mbv program on key aspects of mental health and well-being; specifically, body image and disordered eating symptoms, identity and agency, social and self-constructs, physical health and mood at three time points over the course of the 10-week program, which will be offered remotely in response to the COVID-19 pandemic. Students will be recruited from high schools and will be randomized to receive the mbv program or an assessment-only control group.

DETAILED DESCRIPTION:
Eating disorders have the highest mortality rate of any psychiatric condition and are the second leading cause of mental health disability among young women. Given that eating disorders have their peak onset during adolescence (ages 16-19), prevention efforts among adolescent women are critical in order to avert the onset of these chronic and disabling disorders. The mbv program targets body image and appearance related pressures, awareness of body sensations, and agency and community building skills. The program consists of 10 weekly sessions and is delivered by peer facilitators. This study will implement and evaluate the mbv program at the high school level in order to examine the extent to which the program influences young women's mental health and well-being, particularly related to eating disorder risk factors and symptoms.

Utilizing a randomized controlled trial, the study seeks to address the following aims:

1. To examine the impact of the mbv program on key aspects of mental health and well-being; specifically, body image and disordered eating symptoms, identity and agency, social and self- constructs, physical health and mood among participating high school women.
2. To explore young women's experiences of participating in the program, including strengths and limitations and perspectives on specific activities.

ELIGIBILITY:
Inclusion Criteria:

* High school women, grades 9-12

Exclusion Criteria:

* Prior participation in the Body Project or mind. body. voice. RCT

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 170 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Body Appreciation Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of body appreciation (scale 1-5 with higher scores indicating higher levels of appreciation)
Change in Engaged Living Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of values-based living (scale 1-5 with higher scores indicating higher levels of living based on values)
Change in Multidimensional Assessment of Interoceptive Awareness | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of somatic awareness (scale 1-5 with higher scores indicating higher levels of somatic awareness)
Change in Social Contribution Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of sense of contributing to society (scale 1-5 with higher scores indicating higher levels of contribution)
Change in Sociocultural Pressures Around Appearance | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of sociocultural pressures related to appearance (scale 1-5 with higher scores indicating higher levels of pressure)
Change in Internalization of Media Appearance Ideals | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of internalized appearance ideals in the media (scale 1-5 with higher scores indicating higher levels of internalization)
Change in Ideal Body Stereotype Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of internalization of ideal body stereotypes (scale 1-5 with higher scores indicating higher levels of internalization)
Change in Self-Compassion Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of compassion for oneself (scale 1-5 with higher scores indicating higher levels of self-compassion)
Change in Group Belonging Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of sense of anticipated (baseline) and experienced (follow-up) belonging with intervention program group (scale 1-7 with higher scores indicating higher levels of belonging)
Change in Peer Influence on Appearance Concerns | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of influence of peers on appearance concerns (scale 1-5 with higher scores indicating higher levels of peer influence)
Change in Dieting Behavior and Restraint | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of dieting behavior and restricted eating (scale 1-5 with higher scores indicating higher levels of dieting and restriction)
Change in Body Dissatisfaction Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of body dissatisfaction (scale 1-5 with higher scores indicating higher levels of dissatisfaction
Change in Objectified Body Consciousness Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of body monitoring and surveillance (scale 1-5 with higher scores indicating higher levels of body surveillance)
Change in Self-Liking Scale/Self-Competence Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of how much one likes oneself and considers oneself competent (scale 1-5 with higher scores indicating higher levels of self-liking and self-competence
Change in Self-Efficacy Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of effectiveness in handling challenges and achieving goals (scale 1-5 with higher scores indicating higher levels of self-efficacy)
Change in Belonging Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of general sense of belonging (scale 1-5 with higher scores indicating higher levels of belonging)
Change in Proactive Coping Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of ability to succeed (scale 1-5 with higher scores indicating higher levels of proactive coping)

SECONDARY OUTCOMES:
Change in Eating Attitudes Test 26 | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of disordered eating behaviors (scale 1-6 with higher scores indicating higher levels of disordered eating)
Change in School Engagement and Belonging | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of engagement with schoolwork and belonging in school (scale 1-5 with higher scores indicating higher levels of engagement and belonging)
Change in School Grades and Attendance | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of grades and attendance
Change in Physical Health Questionnaire | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of health outcomes such as sleep and physical symptoms (scale 1-7 with higher scores indicating higher levels of health symptoms)
Change in Positive and Negative Affect Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of positive and negative affect (scale 1-6 with higher scores indicating higher affect levels)
Change in Patient Health Questionnaire A | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of depression (scale 1-4 with higher scores indicating higher levels of depression)
Change in UCLA Loneliness Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of loneliness (scale 1-4 with higher scores indicating higher levels of loneliness)
Change in Humanitarian Egalitarian Scale | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of agreement with humanitarian and egalitarian values (scale 1-5 with higher scores indicating higher levels of agreement)
Change in Generalized Anxiety Disorder 7 | Baseline, midway (5 weeks after baseline), post-intervention (10 weeks after baseline)
  Self-report measure of anxiety (scale 1-4 with higher scores indicating higher levels of anxiety)
Change in COVID-19 impact | Baseline, midway, post-intervention (10 weeks after baseline)
  Self-report measure of COVID-19 negative and positive life impact

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States